CLINICAL TRIAL: NCT02301962
Title: An Open Label, Multicenter, Non-Comparative, Phase IV Study of Panitumumab to Characterize Its Safety, Tolerability and Activity in Indian Subjects With Previously Treated Wild-Type RAS (KRAS and NRAS), Metastatic Colorectal Cancer
Brief Title: Phase IV Panitumumab Study in Indian Subjects With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRL-INDG02-PAN/2018
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Cancer
Keywords: panitumumab; previously treated; metastatic colorectal cancer; fully human antibody; wild-type KRAS and wild-type NRAS
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab arm (Experimental): Subjects will receive panitumumab 6 mg/kg intravenously as monotherapy every 14 days until disease progression, intolerability, withdrawal of consent, or death.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Panitumumab is available as a concentrate for solution for infusion (sterile concentrate). It is a colorless solution that may contain, translucent to white, visible amorphous, proteinaceous panitumumab particles. Each milliliter (mL) of concentrate contains 20 mg panitumumab. Each vial contains 100 mg of panitumumab in 5 mL.

SUMMARY:
This is an open label, multicenter, non-comparative, phase IV study of panitumumab monotherapy in Indian subjects with previously treated, wild-type Kirsten rat sarcoma viral oncogene homolog (KRAS) and wild-type Neuroblastoma rat sarcoma viral (v-ras) oncogene homolog (NRAS), metastatic colorectal cancer. This study is designed to fulfil the requirement of the Indian regulatory authority to characterize the safety and tolerability of panitumumab when administered to Indian subjects with wild-type KRAS and wild-type NRAS metastatic colorectal cancer. Approximately 58 Indian subjects with previously treated wild-type KRAS and wild-type NRAS, metastatic colorectal cancer will be enrolled in order to achieve the target enrollment of 50 evaluable subjects who have received at least one dose of panitumumab. Subjects will receive panitumumab 6 milligram/kilogram (mg/kg) intravenously every 14 days until disease progression, intolerability, withdrawal of consent, or death. All subjects will be followed at 4 weeks and 8 weeks after the last administration of panitumumab, unless the treatment was discontinued due to withdrawal of consent or death of the subject.

DETAILED DESCRIPTION:
This is an open label, multicenter, non-comparative, phase IV study of panitumumab monotherapy in Indian subjects with previously treated, wild-type Kirsten rat sarcoma viral oncogene homolog (KRAS) and wild-type Neuroblastoma rat sarcoma viral (v-ras) oncogene homolog (NRAS), metastatic colorectal cancer. This study is designed to fulfil the requirement of the Indian regulatory authority to characterize the safety and tolerability of panitumumab when administered to Indian subjects with wild-type KRAS and wild-type NRAS metastatic colorectal cancer. Approximately 58 Indian subjects with previously treated wild-type KRAS and wild-type NRAS, metastatic colorectal cancer will be enrolled in order to achieve the target enrollment of 50 evaluable subjects who have received at least one dose of panitumumab. Subjects will receive panitumumab 6 milligram/kilogram (mg/kg) intravenously every 14 days until disease progression, intolerability, withdrawal of consent, or death. All subjects will be followed at 4 weeks and 8 weeks after the last administration of panitumumab, unless the treatment was discontinued due to withdrawal of consent or death of the subject.

All adverse events occurring from signing of informed consent form until 8 weeks after last dose of panitumumab will be recorded. All Serious Adverse Events (SAE) considered related to panitumumab by the investigator or the sponsor will be followed until the event resolves, or is considered stable or until the subject is lost to follow-up or withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally acceptable representative has provided informed consent.
* Male or female >=18 years of age.
* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the colon or rectum.

Metastatic disease.

* Wild-type KRAS (without mutation in exon 2 [codons 12 and 13], exon 3 [codons 59 and 61], and exon 4 [codons 117 and 146]) and wild-type NRAS (without mutation in exon 2 [codons 12 and 13], exon 3 [codons 59 and 61], and exon 4 [codons 117 and 146]) tumor status.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Measurable or non-measurable disease per RECIST Version 1.1.
* Must have failed after fluoropyrimidine-, oxaliplatin-, and irinotecan-containing chemotherapy regimens for metastatic disease. Failure is defined as either disease progression (clinical or radiological) or intolerance to the regimen. Metastatic relapse within 6 months after completing adjuvant chemotherapy (with either an irinotecan or oxaliplatin containing regimen) will also be considered as treatment failure of a prior regimen for metastatic disease. Laboratory: Adequate baseline organ function defined by (<=7 days prior to first dose of study treatment).
* Hematologic function, as follows: Absolute neutrophil count (ANC) >=1.5 x 10^9/Liter (L), Platelet count >=75 x 10^9/L, Hemoglobin >=8.0 gram/deciliter (g/dL).
* Renal function, as follows: Creatinine <=1.5 x upper limit of normal (ULN).
* Hepatic function, as follows: Aspartate aminotransferase (AST) <=3 x ULN, Alanine aminotransferase (ALT) <=3 x ULN, Total Bilirubin <=1.5 x ULN.
* Metabolic function, as follows: Serum Magnesium within normal limits. Serum Calcium within normal limits. Serum Potassium within normal limits.
* All prior treatment related toxicities common terminology criteria for adverse events (CTCAE) version 4.03 <=Grade 1 at the time of enrollment.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use adequate contraception, during the study and for 2 months following the last dose of study treatment. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use adequate contraception, from time of signing informed consent until 5 months after the last dose of study treatment.

Exclusion Criteria:

* History or known presence of central nervous system metastases.
* History of another malignancy except: Malignancy treated with curative intent and with no known active disease present for >=5 years prior to enrolment and felt to be at low risk for recurrence by the treating physician; Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease; Adequately treated cervical carcinoma in situ without evidence of disease; Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to panitumumab or excipients that contraindicates their participation.
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (e.g., panitumumab or cetuximab) or treatment with small molecule EGFr inhibitors (e.g., gefitinib, erlotinib, lapatinib).
* Antitumor therapy (e.g., chemotherapy, hormonal therapy, immunotherapy, antibody therapy, radiotherapy), or investigational agent or therapy <=30 days before first dose of study treatment or not recovered from any acute toxicity.
* Other investigational procedure <=30 days before study entry.
* History of interstitial lung disease (ILD) e.g., interstitial pneumonitis, pulmonary fibrosis or evidence of ILD on baseline chest computer tomography.
* Subject previously enrolled to this study.
* History of keratitis, ulcerative keratitis or severe dry eye.
* Major surgery (e.g., requiring general anesthesia) <=30 days before first dose of study treatment. Subjects must have recovered from any surgery related toxicities.
* Minor surgical procedure (e.g., open biopsy) <=7 days before first dose of study treatment, or not yet recovered from prior minor surgery Note: uncomplicated placement of vascular access device, fine needle aspiration, thoracocentesis or paracentesis >=3 days prior to first dose of study treatment is acceptable.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) <=6 months prior to enrolment.
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with the study participation or investigational product administration, compliance with the study procedures or may interfere with the interpretation of the results.
* Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic event <=30 days before first dose of study treatment. If on anticoagulation, subject must be on stable therapeutic dose prior to first dose of study treatment.
* Subject who is pregnant or breast feeding, or planning to become pregnant during treatment and within 2 months after the discontinuation of study treatment.
* Known positive test(s) for human immunodeficiency virus infection (testing is not required in the absence of clinical suspicion).
* Active infection requiring systemic treatment or any uncontrolled infection <=14 days prior to first dose of study treatment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures or is unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-07-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse event. | 8 months (average duration).
  Adverse events including medically significant laboratory changes- incidence, severity, causality and outcome will be collected from the signing of informed consent form until 8 weeks following discontinuation of study treatment due to disease progression, intolerability, withdrawal of consent or death.

SECONDARY OUTCOMES:
Progression free survival. | Every 8 weeks (assessed up to average of 6 months)
  Progression free survival is defined as the interval between the treatment start date and the earliest date of disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or death due to any cause.
Overall Response Rate. | Every 8 weeks (assessed up to average of 6 months).
  Overall response rate is defined as the percentage of subjects with either a complete response (CR) or partial response (PR) at anytime as per RECIST version 1.1. Where CR is disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline).
Duration of response. | Every 8 weeks (assessed up to average of 6 months).
  Duration of response is defined as the time from initial response (CR or PR) to date of disease progression per RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lalit Lakhwani, MD, Study Director — Dr. Reddys Laboratories Limited
Locations (10):
- India (10):
  - DRL Investigational Site, Vijayawada, Andhra Pradesh
  - DRL Investigational Site, Mumbai, Maharashtra
  - DRL Investigational Site, Nagpur, Maharashtra
  - DRL Investigational Site, Nashik, Maharashtra
  - DRL Investigational Site, Ludhiana, Punjab
  - DRL Investigational Site, Jaipur, Rajasthan
  - DRL Investigational Site, Madurai, Tamil Nadu
  - DRL Investigational Site, Hyderabad, Telangana
  - DRL Investigational Site, Kolkata, West Bengal
  - DRL Investigational Site, New Delhi